CLINICAL TRIAL: NCT04614038
Title: Non-interventional, Prospective, Single-blinded, Observational, Multicenter, Cohort, Clinical Study to Evaluate DETEC® pH Device as a Prognostic Tool in the Identification of Non-healing Chronic Wounds
Brief Title: DETEC® pH Point of Care Wound Diagnostic Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Progenitec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DETEC 001
Record Dates: First submitted 2020-10-22; First posted 2020-11-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer; Wound, Non-Healed
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: DETEC® pH — DETEC® pH is a disposable diagnostic device that is used to indicate the alkalinity of the wound by testing wound exudate adsorbed onto wound dressing.

SUMMARY:
The purpose of this study is to determine the relationship between wound alkalinity and the non-healing status of chronic ulcer wounds. It is hypothesized that wounds with an alkaline environment as indicated by DETEC pH will have a high chance of not healing over 12 weeks of wound care.

DETAILED DESCRIPTION:
Chronic wounds fail to progress through normal wound healing phases in a timely manner which makes them non-healing over time. The inability to identify a slowly healing or non-healing wound early on can be detrimental to the patient's well-being. Currently, determination of non-healing wounds is based on the clinician's visual observation of wound size changes for 4 weeks. Many early studies have documented that chronic, non-healing, or infected wounds often reside in an alkaline state (pH > 7.2) while healing wounds are habitually associated with a non-alkaline and even acidic environment.

To reliably and continuously monitor wound alkalinity objectively, a portable, disposable, non-invasive, and non-contact device - DETEC® pH - was developed to indirectly assess the alkalinity of wounds by analyzing the wound exudate adsorbed on to freshly discarded wound dressings during the participants' routine follow-up visit. A follow-up visit and 7-21 days after the initial wound diagnosis and care, subjects will be screened and enrolled in this investigation based on the inclusion and exclusion criteria. Their wound dressings will be tested using the device. The device outputs and wound conditions will be recorded. The subjects' wounds will be managed using standard care by the provider at each visit. The device output will not be used to inform the treatment decision in this study.

At 12 weeks after initial wound diagnosis, the subjects will be required to present themselves for a follow-up/end of study wound healing status assessment.

The device outputs will then be compared to the clinical healing status of the wounds (healed or not healed) at week 12. For the study, a healed wound is defined as one that has achieved complete wound closure that is defined as skin re-epithelialization without drainage or dressing requirements (100% of the wound is covered and the surface is intact), as assessed by the treating clinician.

ELIGIBILITY:
Inclusion Criteria:

* Adult (21 years), male or female, inpatient/outpatient, presenting with a wound
* Chronic wound open for at least 30 days, including (Diabetic foot ulcers (DFU), Wagner grade 1 to 3), (Pressure ulcers, stage 2 to 4), (Venous leg ulcers (VLU), confirmed by venous duplex/Doppler),
* For wounds on a lower extremity (i.e. DFU, VLU) an ankle-brachial index (ABI) of greater than 0.6 for the affected leg to ensure ischemia will not impact healing
* For diabetic foot ulcers - confirmed type 1 or type 2 diabetes mellitus with a hemoglobin A1C less than 10 percentage

Exclusion Criteria:

* History of autoimmune disease/ acquired immunodeficiency syndrome/Hepatitis
* Require treatment for primary or metastatic malignancy
* Any contra-indication to routine wound care and/or monitoring
* Women who are pregnant, lactating, or of childbearing potential and currently not taking adequate birth control
* Scheduled for or likely to have significant surgical intervention to the studied wound (e.g. skin graft or flap, amputation) during the study period.
* With a life expectancy of fewer than 6 months
* Participation (less than 30 days prior to baseline) in an interventional trial which could have a potential effect on the study outcome, as determined by the Investigator
* Patients with a dry dressing

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have shown no significant progress toward healing in 30 days and thus been diagnosed with chronic wounds.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-healing status based on change in wound area over 12 weeks | 12 weeks from enrollment
  The primary endpoint is non-healing wounds (that do not have 100 percent wound closure) at the end of 12 weeks

SECONDARY OUTCOMES:
Effect of various patient biometry and wound conditions on non-healing status based on change in wound area over 12 weeks | 12 weeks from enrollment
  The secondary effectiveness endpoint is healing or non-healing wounds over 12 weeks based on subject's age, race, initial wound size, wound location, wound type, clinical sites and presence or absence of infection

CONTACTS AND LOCATIONS:
Overall Officials: Wenjing Hu, Ph.D., Principal Investigator — Progenitec Inc.
Locations (2):
- United States (2):
  - Northwell Health Comprehensive Wound Healing Center, Lake Success, New York
  - Complex Healthcare Solutions, Arlington, Texas